CLINICAL TRIAL: NCT02523950
Title: Evaluation of Staged and Combined Phacoemulsification With Intraocular Lens (IOL) Implantation and Descemet Membrane Endothelial Keratoplasty (DMEK) for Cataract Patients With Corneal Endothelial Dysfunction
Brief Title: Staged and Combined Surgery for Cataract Patients With Corneal Endothelial Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haotian Lin (Other)
Responsible Party: Sponsor-Investigator, Haotian Lin, M.D., Ph.D., Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015MEKY047
Record Dates: First submitted 2015-07-07; First posted 2015-08-14 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Cataract; Corneal Endothelial Keratopathy; Phacoemulfisication+IOL Implantation; Endothelial Keratopathy
MeSH Terms: conditions — Cataract | interventions — Lenses, Intraocular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Staged group (Active Comparator): Procedure/Surgery: Phacoemulsification + IOL implantation is performed in the first stage and DMEK is performed secondarily.
  Interventions: Procedure: Staged phacoemulsification and DMEK; Device: Intraocular lens (IOL) implantation
- Combined group (Active Comparator): Procedure/Surgery: Phacoemulsification + IOL implantation and DMEK are performed simultaneously.
  Interventions: Procedure: Combined phacoemulsification and DMEK; Device: Intraocular lens (IOL) implantation

INTERVENTIONS:
Procedure: Staged phacoemulsification and DMEK — Stage 1. Phacoemulsification is performed individually. During phacoemulsification, viscoelastic materials and anterior lens capsule are used to protect corneal endothelial cells.
  Stage 2. DMEK is performed secondarily according to the corneal status of patients.
  Arms: Staged group
Procedure: Combined phacoemulsification and DMEK — Routine phacoemulsification and DMEK are performed simultaneously.
  Arms: Combined group
Device: Intraocular lens (IOL) implantation — After phacoemulsification and removal of all the lens material, a one-piece IOL is implanted into the lens capsule.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of staged and combined phacoemulsification with intraocular lens implantation and Descemet membrane endothelial keratoplasty (DMEK) to treat cataract patients with corneal endothelial dysfunction. Surgical and postoperative complications, visual acuity and corneal endothelial cell density are evaluated.

DETAILED DESCRIPTION:
The prospective, randomized, controlled study involves the enrollment of cataract patients with corneal endothelial dysfunction. All the patients will be randomly assigned with equal probability to the following two groups: 1. Staged group: phacoemulsification + IOL implantation is performed individually and DMEK is performed secondarily according to the corneal status of patients. During cataract surgery, viscoelastic materials and anterior lens capsule are used to protect the compromised corneal endothelium during phacoemulsification. After phacoemulsification and removal of all the lens material, a one-piece foldable IOL is implanted into the lens capsule. 2: Combined group: phacoemulsification + IOL implantation and DMEK is performed simultaneously. Standard procedures of phacoemulsification + IOL implantation are the same as in the staged group.

Patients enrolled into the study will be followed for one year and will have study visits at 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after each surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are older than 18 years.
2. Subjects have corneal endothelial dysfunction combined with cataract.
3. Subjects have mild to moderate cortical and/or nuclear cataract.
4. Subjects are able and willing to provide informed consent.

Exclusion Criteria:

1. Subjects have corneal stromal opacity and/or neovascularization.
2. Subjects have other intraocular disease that disturbs visual rehabilitation.
3. Subjects have corneal infection, perforation or scarring.
4. Subjects are pregnant.
5. Subjects have concurrent disease that could confound the response to therapy.
6. Subjects are unlikely to comply with the protocol or likely to be lost to follow-up.
7. Subjects have known hypersensitivity or intolerance to the proposed therapy.
8. Subjects use concomitant therapy that affects either tear function or ocular surface integrity.
9. Subjects have had surgical or other manipulation of the eye that could confound the outcome parameters or interfere with the mechanism of action of the proposed intervention to be studied.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual acuity measured by Snellen chart | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery
Change from baseline in central corneal thickness measured by anterior segment OCT | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery
Change from baseline in endothelial cell density measured by corneal specular microscopy | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery

SECONDARY OUTCOMES:
Change from baseline in endothelial graft attachment measured by anterior segment OCT | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery
Change from baseline in corneal transparency measured by slit-lamp microscopy | 1 day, 1 week, 2 weeks, 1 month, 3 months, 6 months and 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, M.D., Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Wang Y, Xia Y, Zeng M, Liu X, Luo L, Chen B, Liu Y, Liu Y. Torsional ultrasound efficiency under different vacuum levels in different degrees of nuclear cataract. J Cataract Refract Surg. 2009 Nov;35(11):1941-5. doi: 10.1016/j.jcrs.2009.05.055. PMID 19878827
- [Background] Huang T, Wang Y, Ji J, Gao N, Chen J. Deep lamellar endothelial keratoplasty for iridocorneal endothelial syndrome in phakic eyes. Arch Ophthalmol. 2009 Jan;127(1):33-6. doi: 10.1001/archophthalmol.2008.537. PMID 19139335
- [Background] Luo L, Lin H, He M, Congdon N, Yang Y, Liu Y. Clinical evaluation of three incision size-dependent phacoemulsification systems. Am J Ophthalmol. 2012 May;153(5):831-839.e2. doi: 10.1016/j.ajo.2011.10.034. Epub 2012 Feb 4. PMID 22310081
- [Background] Xia Y, Liu X, Luo L, Zeng Y, Cai X, Zeng M, Liu Y. Early changes in clear cornea incision after phacoemulsification: an anterior segment optical coherence tomography study. Acta Ophthalmol. 2009 Nov;87(7):764-8. doi: 10.1111/j.1755-3768.2008.01333.x. Epub 2009 Jun 22. PMID 19548882
- See also: Zhongshan Ophthalmic Center website — http://www.gzzoc.com